CLINICAL TRIAL: NCT05725811
Title: Immediate Effects of Myofascial Release on the Quadriceps or Hamstrings on Active Cervical Flexion and Extension Range of Motion
Brief Title: Immediate Effects of Myofascial Release on the Quadriceps or Hamstrings on Active Cervical Range of Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Fernando Pessoa (Other)
Responsible Party: Principal Investigator, Ricardo Cardoso, Professor, University Fernando Pessoa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ESS/FSA-206/22-2
Record Dates: First submitted 2023-01-25; First posted 2023-02-13 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group 1 (Active Comparator): A myofascial release technique will be performed using a foam roller (Blackroll Standard, 30 x 15 cm) on the dominant lower limb.
  For the IG 1, the technique will be applied to the hamstrings muscles. In this group, participants will sit on the floor on a mat with the roller under their thighs. Their hands will be placed on the floor with their fingers pointing downwards. The foam roller will be in contact with the muscle being tested and the patient will exert a load until they feel a slight pain. In this way, the patient performs a self-massage in the direction of the muscle fibers. The limb that will not be tested will function as a lever, it will remain bent to the side, which will allow the simple realization of the glide.
  A cycle of the procedure will be defined as a proximal to distal rolling movement, so the frequency in this study will be 25 cycles per minute measured with a metronome from a mobile application (Smart Metronome & Tuner v.11.8 IOS).
  Interventions: Other: Dynamic foam rolling
- Intervention group 2 (Active Comparator): A myofascial release technique will be performed using a foam roller (Blackroll Standard, 30 x 15 cm) on the dominant lower limb.
  The IG 2 will perform the same technique on a different muscle group: the quadriceps. In this way, the positioning will be different, the participants will be in the prone position, in a plank position, leaning on the forearms, the body well aligned and the studied lower limb well stretched. However, the participant will also perform a self-massage in the direction of the muscle fibers until they feel slight pain. The duration of the procedure will be set at 4 minutes in this study; 3 rounds of 1 minute (30 s rest).
  A cycle of the procedure will be defined as a proximal to distal rolling movement, so the frequency in this study will be 25 cycles per minute measured with a metronome from a mobile application (Smart Metronome & Tuner v.11.8 IOS).
  Interventions: Other: Dynamic foam rolling
- Control group (No Intervention): The participants will remain at rest in a chair for 4 minutes.

INTERVENTIONS:
Other: Dynamic foam rolling — The foam roller will be in contact with the muscle being tested and the patient will exert a load until they feel a slight pain. In this way, the patient performs a self-massage in the direction of the muscle fibers.
  Arms: Intervention group 1; Intervention group 2

SUMMARY:
The purpose of this study is to verify the immediate effects of quadriceps or hamstring myofascial release on the active cervical flexion and extension range of motion.

DETAILED DESCRIPTION:
After completing the questionnaire, 60 healthy college students will be randomly divided into three groups named Intervention Group 1 (IG 1) (n=20), Intervention Group 2 (IG 2) (n=20) and Control Group (CG) (n=20). In the first assessment (M0), the cervical flexion and extension range of motion will be measured with a goniometer. The myofascial release technique (foam roller) will be applied on the hamstrings (IG 1) or quadriceps (IG 2) of the dominant lower limb for 4 minutes (3 series of 1 minute with 30s rest). Participants in the control group will remain at rest sitting in a chair for 4 minutes.

Immediately after the intervention/control, both groups will be assessed, again (M1).

ELIGIBILITY:
Inclusion Criteria:

* Healthy university students of both genders with normal mobility of the joints.

Exclusion Criteria:

* Deformities in the lower quadrant region of the body;
* Complaints in this region in the last 6 months;
* Surgical procedures or musculoskeletal, cardiac, renal, metabolic, neurological and or oncological pathologies
* Pregnant women
* Ingestion of non-steroidal anti-inflammatory drugs or consumption of any type of narcotic drugs and participants who have drunk alcohol in the last 12 hours.

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Change of active cervical range of motion in flexion and extension. | Change from Baseline (M0) to Immediately after intervention or control (M1)
  Data will be collected in two moments: baseline (M0) and after the intervention/control (M1). Participants will be asked to sit with their spine straight against the back of the chair. The ankles, knees and hips of the subjects will be positioned at right angles and the arms crossed over the chest to minimize thoracic movements.
  The position of the goniometer (GIMA, 37.5 x 6.5 x 0.5 cm) will be as follows: the fixed point at the level of the external acoustic meatus, and the mobile arm at the level of the base of the nose (initial position: 90°). The fixed arm will be immobile, parallel to the ear and perpendicular to the ground. Prior to the test, each participant will have performed both movements until the final sensation is reached in order to increase the fluidity of the test. Thus, the first movement asked of the patient will be a flexion followed by an extension (the examiner will take the average of three measurements).

CONTACTS AND LOCATIONS:
Locations (1):
- Ricardo Cardoso, Porto, Portugal